CLINICAL TRIAL: NCT04469192
Title: The Efficacy of Cryotherapy in Pregnancy Related Pelvic Girdle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Colleen M. Fitzgerald, MD, MS, MD, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 212358
Record Dates: First submitted 2020-06-16; First posted 2020-07-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Cryotherapy; Educational Status

STUDY DESIGN:
Intervention Model Description: Study participants will then be randomized to cryotherapy + education vs. education alone. The education portion will consist of a handout that will be provided to each patient describing specific exercises. These exercises include descriptive information along with pictures on ways to improve posture and protect the lower back in pregnancy good posture.
  Those randomized to the intervention group will receive a 20-minute topical cryotherapy treatment (using Medline Deluxe Cold Pack) at this initial visit where they will be monitored for any adverse response as well as for any immediate change to the NPRS and PGQ. The participant will place the icepack over the low back region and the sacrum if the pain is bilateral. If the pain is unilateral will place the icepack over just that side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cryotherapy + education (Experimental): intervention group will receive a 20-minute topical cryotherapy treatment (using Medline Deluxe Cold Pack) The education portion will consist of a handout that will be provided to each patient describing specific exercises. These exercises include descriptive information along with pictures on ways to improve posture and protect the lower back in pregnancy good posture
  Interventions: Other: Cryotherapy; Other: Education
- education alone (Active Comparator): The education portion will consist of a handout that will be provided to each patient describing specific exercises. These exercises include descriptive information along with pictures on ways to improve posture and protect the lower back in pregnancy good posture
  Interventions: Other: Education

INTERVENTIONS:
Other: Cryotherapy — intervention group will receive a 20-minute topical cryotherapy treatment (using Medline Deluxe Cold Pack) The education portion will consist of a handout that will be provided to each patient describing specific exercises. These exercises include descriptive information along with pictures on ways to improve posture and protect the lower back in pregnancy good posture
  Arms: cryotherapy + education
Other: Education — The education portion will consist of a handout that will be provided to each patient describing specific exercises. These exercises include descriptive information along with pictures on ways to improve posture and protect the lower back in pregnancy good posture

SUMMARY:
The findings from this project may result in pain reduction and improved mobility in pregnant women with pelvic girdle pain in their second and third trimester.

DETAILED DESCRIPTION:
The primary objective of this unblinded randomized controlled trial is to determine whether superficial cryotherapy results in improved Numeric Pain Rating Scale (NPRS) scores among pregnant women with posterior pelvic girdle pain. The investigators hypothesize that superficial cryotherapy, in addition to receipt of an educational pamphlet, will result in improved NPRS scores compared to receipt of an educational pamphlet alone.

This study will include English-speaking pregnant women presenting to Loyola University Medical Center obstetrics or rehabilitation clinics in their second or third trimester with posterior pelvic girdle pain, defined as an NPRS score > 2 onset within the past 3 months and pain experienced between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joints (SIJ). The pain may radiate in the posterior thigh and can also occur in conjunction with/or separately in the [pubic] symphysis. NPRS scores will be measured as a continuous, numerical integer ranging from a value of 0 (No pain) to a value of 10 (Worst possible pain).

ELIGIBILITY:
Inclusion Criteria:

* English speaking pregnant women presenting in their second or third trimester with acute posterior PGP (occurring within the last 3 months). Trimester will be determined from the date of last menses or ultrasound date.
* Current VAS pain score between 2-4
* Written informed consent

Exclusion Criteria:

* Non-English speaking pregnant women <18 or >50 years old
* Women presenting with low back pain, or posterior pelvic pain in the first trimester (<13 weeks gestation).
* Women with acute low back pain in 2nd and 3rd trimester
* Women with anterior pelvic girdle pain (pubic symphysis) alone
* Chronic low back pain (current or past history, defined as > 6 weeks of low back pain)
* History of lumbar or pelvic fracture; degenerative disc disease; neoplasm; inflammatory disease; active urogenital infection or active gastrointestinal illness; previous surgery of the lumbar spine, pelvic girdle, hip joint or femur
* History or signs of radiculopathy or other systemic neurologic disease
* Narcotic medication use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change in pelvic girdle pain using the Numeric Pain Rating Scale | On day 6
  The change in the Numeric Pain Rating Scale (NPRS) from baseline to day 6 (i.e., the delta value of NPRS) will be compared between the two groups. NPRS scores range from 0 (no pain) to 10 (worst possible pain).
Change in pelvic girdle pain using the Pelvic Girdle Questionnaire | On day 6
  The change in the the Pelvic Girdle Questionnaire (PGQ) from baseline to day 6 (i.e., the delta value of PGQ) will be compared between the two groups. The PGQ measures problems with carrying out daily activities and ranges from 0 (no problem at all) to 100 (experiences problems to a large extent).

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Fitzgwerald, MD, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States